CLINICAL TRIAL: NCT01057446
Title: Prospective Randomized Comparison of Oral Sodium Phosphate and Sennoside A+B Calcium Lavage for Colonoscopy Preparation
Brief Title: Comparison of Oral Sodium Phosphate and Sennoside A+B Calcium Lavage for Colonoscopy Preparation
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Manuk Manukyan MD, Maltepe University
Other Study IDs: mütf
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2009-11

CONDITIONS: Colonoscopy
Keywords: Colonoscopy preparation; sennoside; sodium phosphate; the aim is to assess the bowel cleansing effects of two different agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the investigators study is to assess the bowel cleansing effects of two different agents and to compare their safety of application, ease of usage and effects on serum electrolytes.

DETAILED DESCRIPTION:
Colorectal cancer is a leading cause of death from cancer. Because colonic cancer begins as a small adenoma that , evolves into carcinoma over a decade or more pre-emptive colonoscopic polypectomy can prevent this malignancy. For a good colonoscopic examination ideally the colon should be cleansed of all fecal material because poor bowel preparation before colonoscopy often leads to inability to reach the cecum or poor visualization of the mucosa . Thus , pathology may be missed, repeat examinations may be scheduled at earlier intervals than planned and the procedure is more difficult and time consuming. In addition , poor bowel preparation can increase the risk of significant complications. Perforations resulting from maneuvers has greater consequences in the setting of inadequate bowel preparation.

In the past two decades , various bowel preparation methods have been proposed including castor oil, anthraquinones, phenolphtalein and magnesium citrate, in combination with low residue diet4-7. Along these agents , cleansing enemas formed the traditional bowel preparation. Oral sodium phosphate (Fleet Phospo-soda, C.B Fleet Co, Inc., Lynchburg, Va.)(NaP) a preparation containing dibasic and monobasic sodium phosphate was proven to be cost effective and has since been used worldwide8,9. NaP osmotically draws plasma water into the bowel lumen to promote bowel cleansing. NaP must be accompanied by significant oral fluid to prevent dehydration. Patients with compromised renal function, dehydration, hypercalcemia or hypertension with the use of angiotensin converting enzyme inhibitors have experienced phosphate nephropathy after use of oral NaP solutions.

Senna laxatives containing sennosides activated by colonic bacteria have a direct effect on intestinal mucosa increasing the rate of colonic motility , enhancing colonic transit, and inhibiting water and electrolyte secretion10. Sennosides may result in hypokalemia and atonic colon.

The aim of our study is to assess the bowel cleansing effects of two different agents and to compare their safety of application, ease of usage and effects on serum electrolytes.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring diagnostic outpatient colonoscopy.
* Over the age of 18 and giving informed consent by their will.

Exclusion Criteria:

* Patients unable to give informed consent
* Those younger than 18 years old
* Those with a known history of chronic renal failure
* Pregnant women and those with a known history of bowel resection were excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ninety-nine patients requiring diagnostic outpatient colonoscopy were prospectively recruited for the study and randomized by internet based Easy sample random numbers software program to two arms of sodium phosphate versus Sennosid A+B calcium preparation.
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
Colonic cleansing was evaluated by using the amount and consistency of stool remained in the colonic segment

REFERENCES:
- [Derived] Manukyan MN, Tolan K, Severge U, Attaallah W, Kebudi A, Cingi A. Prospective randomized comparison of oral sodium phosphate and sennoside A+B calcium lavage for colonoscopy preparation. Surg Laparosc Endosc Percutan Tech. 2011 Apr;21(2):90-3. doi: 10.1097/SLE.0b013e31820e8793. PMID 21471799